CLINICAL TRIAL: NCT03665558
Title: Effect of DDD Pacing Titrated by Stepwise Changing of AVD on Aortic dP/dt
Brief Title: Effect of Pacing on Aortic dP/dt Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Murat Sezer, Clinical Professor, Istanbul University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 843-1075
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-09

CONDITIONS: Aortic Diseases
Keywords: Ventricular contractility; Pacing; Ventricular dP/dt; Aortic dP/dt
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aortic dP/dt in sinus rhythm (No Intervention): Left ventricular and aortic dP/dt values were recorded at baseline condition while patients are on sinus rhythm.
- Aortic dP/dt during DDD pacing (Active Comparator): Patients will be their own control. Aortic and ventricular pressures will be recorded under temporary DDD pacing again and these data collected at every pacing steps will be compared to the pressures recorded at baseline condition.
  Interventions: Device: Temporary DDD pacing

INTERVENTIONS:
Device: Temporary DDD pacing — Measurements will be performed in patients otherwise undergoing invasive catheterization procedure. Baseline ventricular and aortic hemodynamic parameters (continuous pressure recordings) will be recorded. Thereafter, DDD pacing with stepwise changing of the AV delay will be performed. During each pacing steps left ventricular and aortic pressures at different aortic levels will be continuously recorded. From these hemodynamic data, left ventricular and aortic dP/dt values will be calculated off line.
  Arms: Aortic dP/dt during DDD pacing

SUMMARY:
The maximum value of rate of left ventricular pressure increase, denoted by left ventricular peak dP/dt value (dP/dt max), corresponds to the highest point on the curve of first derivative of ventricular pressure curve with respect to time. It is one of the important systolic performance parameters, which is primarily determined by ventricular contractility, and emerges in isovolumetric contraction phase when aortic valves are closed. Thus it is not influenced by parameters beyond ventricle such as aortic valve area, aortic elastance and peripheral resistance. Despite these unique advantageous, the main reason for its limited usage in assessing ventricular systolic performance instead of commonly used ejection fraction is the difficulties in its calculation, which requires incessant intraventricular pressure recordings.

The maximum value of acceleration rate of aortic pressure increase can be named as aortic peak dP/dt. It, likewise, corresponds to the maximum value of first derivative of pressure curve with respect to time.

Since it is one of the principal determining factors of aortic peak dP/dt, changing left ventricular contractility thereby left ventricular peak dP/dt value is expected to change aortic peak dP/dt in the same direction since all other variables being unchanged. Yet to conclude the extent of this association and magnitude of change, measuring these parameters for various contractility levels is necessary. In addition, impact of decreasing left ventricular peak dP/dt by gradually lowering ventricular contractility upon aortic peak dP/dt has not been investigated in previous studies.

In the present study, changes in left ventricular and aortic peak dP/dt values in response to gradual reduction in LV contractility with stepwise changing (decremental shortening) atrio-ventricular delay (AVD) by dual chamber pacing will be investigated in patients without systolic dysfunction.

DETAILED DESCRIPTION:
The maximum value of rate of left ventricular pressure increase, denoted by left ventricular peak dP/dt value (dP/dt max), corresponds to the highest point on the curve of first derivative of ventricular pressure curve with respect to time. It is one of the important systolic performance parameters, which is primarily determined by ventricular contractility, and emerges in isovolumetric contraction phase when aortic valves are closed. Thus it is not influenced by parameters beyond ventricle such as aortic valve area, aortic elastance and peripheral resistance. Despite these unique advantageous, the main reason for its limited usage in assessing ventricular systolic performance instead of commonly used ejection fraction is the difficulties in its calculation, which requires incessant intraventricular pressure recordings.

The maximum value of acceleration rate of aortic pressure increase can be named as aortic peak dP/dt. It, likewise, corresponds to the maximum value of first derivative of pressure curve with respect to time. Unlike left ventricular peak dP/dt, it emerges after aortic valve opens in early systolic ejection phase and thus is influenced by parameters beyond ventricle in addition to left ventricular contractility such as aortic elastance and compliance, vascular resistance, interference of forward and backward propagating pressure waves, stroke volume and its ejection rate (dV/dt). Notably, aortic peak dP/dt can be expected to be one of principal determinants in pressure-related damages in the vascular system. In structures exposed to variable pressures, the extent of damage depends on the magnitude and rate of acceleration of applied pressure in addition to susceptibility of the structures. Whether this mechanism, which has numerous implications from the real world, operates in the organism as well can be exemplified by the pulse pressure, which is an independent risk factor for adverse cardiovascular events apart from systolic and diastolic blood pressure levels. A wide pulse pressure suggests an accelerated rate of pressure increase. Therefore applications lowering left ventricular and aortic peak dP/dt values may open a new therapeutic avenue in management of pressure-related vascular damages such as aortic aneurisms. However, aortic peak dP/dt concept is seldom found a place even in research articles.

Since it is one of the principal determining factors of aortic peak dP/dt, changing left ventricular contractility thereby left ventricular peak dP/dt value is expected to change aortic peak dP/dt in the same direction since all other variables being unchanged. Yet to conclude the extent of this association and magnitude of change, measuring these parameters for various contractility levels is necessary. In this context, it has been demonstrated that narrowing of the QRS complex by cardiac resynchronization therapy (CRT) was shown to increase left ventricular peak dP/dt value. This finding strongly suggests that widening of the QRS complex, on the contrary, will decrease left ventricular peak dP/dt value. However, impact of decreasing left ventricular peak dP/dt by gradually lowering ventricular contractility upon aortic peak dP/dt has not been investigated in previous studies.

In the present study, changes in left ventricular and aortic peak dP/dt values in response to gradual reduction in left ventricular (LV) contractility with stepwise changing (decremental shortening) atrio-ventricular delay (AVD) by dual chamber pacing will be investigated in patients without LV systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

• Normal left ventricular systolic function

Exclusion Criteria:

* Abnormal left ventricular systolic function with ejection fraction < 50%
* Presence of severe coronary artery disease
* Presence of valvular heart disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Changing in aortic dP/dt in response to DDD pacing | At the end of the stepwise pacing procedure completed
  Changing in aortic dP/dt in response to DDD pacing will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sezer M, Atici A, Coskun I, Cizgici Y, Ozcan A, Umman B, Bugra Z, Ozcan I, Hasdemir H, Kocaaga M, Davies JE, Umman S. Reducing Aortic Barotrauma and Vascular Extracellular Matrix Degradation by Pacemaker-Mediated QRS Widening. J Am Heart Assoc. 2020 May 18;9(10):e014804. doi: 10.1161/JAHA.119.014804. Epub 2020 May 11. PMID 32390533